CLINICAL TRIAL: NCT05015374
Title: Effect of Astaxanthin on the Patients With Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB- F(II)-20180054
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-07

CONDITIONS: To Evaluate the Possible Benefit of Astaxanthin on Alzheimer Disease
Keywords: Alzheimer disease; Astaxanthin
MeSH Terms: conditions — Alzheimer Disease | interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Compared the difference of changes in psychometrics between Astaxanthin users and placebo group.
  Interventions: Dietary Supplement: Placebo
- Astaxanthin (Active Comparator): Compared the difference in adverse effects between Astaxanthin users and placebo group.
  Interventions: Dietary Supplement: Astaxanthin

INTERVENTIONS:
Dietary Supplement: Astaxanthin — 350 mg/capsule (2mg Astaxanthin)
  Arms: Astaxanthin
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
This study adapts a randomized, double-blind, placebo-controlled trial, to exam the possible benefit of Astaxanthin on Alzheimer disease. The enrolled Alzheimer patients will take Astaxanthin or placebo for 1 year. We will follow up Mini-Mental State Examination, Cognitive Ability Screening Instrument, Clinical Dementia Rating, and Neuropsychiatric Inventory at the end of the study.

DETAILED DESCRIPTION:
This study aims to examine the benefit of Astaxanthin as adjuvant therapy for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. 60 ≦ age ≦ 90
2. Clinical Dementia Rating Scale = 0.5 or 1
3. Under treatment with donepezil、rivastigmine or galantamine with good medical adherence
4. Get a signed informed consent from the patient or his/her family

Exclusion Criteria:

1. Not using or poor medical adherence to donepezil、rivastigmine or galantamine
2. Combined using memantine or other cerebral perfusion enhancing agent, such as Piracetam, Dihydroergotoxine, Nicergoline etc.
3. New cerebrovascular disease happens during 3-year follow up
4. Mixed type dementia
5. Major psychiatric disease (such as depression, bipolar disorder, schizophrenia) or substance abuser (such as alcohol, illegal drug, hypnotics)
6. Heart failure, end stage renal disease, liver cirrhosis, or other major organ failure
7. Severe hearing impairment results in incomplete survey of neuropsychatric evaluation
8. No informed consent or no regular follow up

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 3 years
  All participants receive MMSE when they are enrolled, and follow up annually for a total of 3 years.
Cognitive Ability Screening Instrument (CASI) | 3 years
  All participants receive CASI when they are enrolled, and follow up annually for a total of 3 years.
Clinical Dementia Rating (CDR) | 3 years
  All participants receive CDR when they are enrolled, and follow up annually for a total of 3 years.
Neuropsychiatric Inventory (NPI) | 3 years
  All participants receive NPI when they are enrolled, and follow up annually for a total of 3 years.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events [safety and tolerability] | 3 years
  Monitor possible adverse effects of Astaxanthin, namely bleeding, anemia, blood sugar, blood pressure, liver and renal functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Will not share individual participant data